CLINICAL TRIAL: NCT06079814
Title: Virtual Reality Application for Pain and Anxiety Reduction During Cystoscopy: A Randomized Controlled Study
Brief Title: Virtual Reality Application for Pain and Anxiety Reduction During Cystoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Seyma Yurtseven, Clinic Nurse, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5312256929
Record Dates: First submitted 2023-10-02; First posted 2023-10-12 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): Patients will wear virtual reality glasses 10 minutes before cystoscopy. The content chosen by the patient (there will be three options) will be watched throughout the procedure.
  Interventions: Other: virtual reality intervention
- control group (No Intervention): Standard procedure.

INTERVENTIONS:
Other: virtual reality intervention — Patients will be shown content through the patient's virtual reality glasses throughout the cystoscopy procedure.
  Arms: experiment group

SUMMARY:
The aim of this research is to conduct a two-group randomized controlled intervention study to determine the effect of virtual reality applications on pain and anxiety during cystoscopy. The study population will consist of patients who have applied to the urology outpatient clinic of a University Hospital for cystoscopy. The study sample will be composed of patients who volunteer to participate in the study and meet the criteria during the planned dates of the research. Data will be collected using a 'Personal Information Form' created by the researcher through a literature review, the 'Visual Analog Scale' (VAS) for assessing pain, and the 'State Anxiety Inventory' (SAI) for assessing anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Being literate,
* Being conscious,
* Ability to understand and speak Turkish and not have hearing or visual impairment,
* Agreeing to participate in the research.

Exclusion Criteria:

* Having a diagnosed psychiatric and mental illness,
* Patients diagnosed with epilepsy (due to the risk of virtual reality glasses triggering epileptic seizures),
* Patients who do not want to continue the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
The effect of virtual reality applications on pain during cystoscopy | 30 minutes after the procedure
  The patient's pain will be assessed using the 'Visual Analog Scale (VAS).' This scale involves marking on a 10 cm vertical or horizontal line, with one end indicating no pain at all and the other end indicating the most severe pain, to assess and measure the level of pain.
The effect of virtual reality applications on anxiety during cystoscopy | 30 minutes after the procedure
  Procedure related anxiety will be assessed using the 'State Anxiety Inventory.' This inventory consists of a total of 20 items and the scoring ranges from 20 to 80 points. The higher the total score obtained from the scale, the higher the level of anxiety experienced by the individual is interpreted.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided